CLINICAL TRIAL: NCT01114620
Title: Immunogenicity and Safety Study of GSK Biologicals' Influenza Vaccine Arepanrix™ (GSK2340274A) in Adults 65 Years of Age or Older
Brief Title: Study of GSK Biologicals' Influenza Vaccine Arepanrix™ in Japanese Adults 65 Years of Age or Older
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 114270
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Influenza
Keywords: elderly; post-marketing; H1N1; Clinical trial; pandemic influenza
MeSH Terms: conditions — Influenza, Human | interventions — arepanrix

ARMS (1):
- Arepanrix Group (Experimental): Healthy Japanese male and female adults, 65 years of age or older, who received one dose of the study vaccine Arepanrix™, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
  Interventions: Biological: Arepanrix™

INTERVENTIONS:
Biological: Arepanrix™ — Intramuscular administration, one dose

SUMMARY:
The purpose of this study is to comply with the post marketing condition to the exceptional approval of Arepanrix™ in Japan and to assess the immunogenicity and safety of GSK Biologicals' H1N1 influenza vaccine healthy Japanese adults 65 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female adults 65 years of age or older at time of vaccination.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Good general health as assessed by medical history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception and for 2 months after study vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* History of previous administration of a pandemic H1N1 vaccine.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence or evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5 °C, or acute symptoms greater than "mild" severity on the scheduled date of vaccination.
* Diagnosed with cancer, or treatment for cancer within three years.

  * Persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
  * Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are accepted and may enrol, but other histologic types of skin cancer are exclusionary.
  * Women who are disease-free three years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enroll.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period. For corticosteroids, this will mean a dose equivalent to 10 mg/day of prednisone or equivalent when administered for > 2 weeks. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within three months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 months of receipt of seasonal influenza vaccination.
* Administration of any vaccines within 30 days before vaccination or planned administration before blood sampling at Day 21 and within 30 days prior to blood sampling at Day 182.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Excessive underweight [Body Mass Index (BMI) < 18.5] or excessive obesity (BMI >= 30).
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.
* Clinically or virologically confirmed influenza infection within 12 months preceding the study start.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2010-11-05 (Actual); Study Completion 2010-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ikematsu H, Tenjinbaru K, Li P, Madan A, Vaughn D. Evaluation of immune response following one dose of an AS03A-adjuvanted H1N1 2009 pandemic influenza vaccine in Japanese adults 65 years of age or older. Hum Vaccin Immunother. 2012 Aug;8(8):1119-25. doi: 10.4161/hv.21081. Epub 2012 Aug 1. PMID 22854661
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arepanrix Group
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.8 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese heritage | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Hemagglutination Inhibition (HI) Antibodies
Description: Seroconversion (SCR) was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 30

2. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: Seroprotection (SPR) was defined as the proportion of subjects with H1N1 reciprocal HI titers equal to or above (≥) 40 against the tested vaccine virus. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 32

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: GMFR, also known as seroconversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Fold change | 10.2 [6.9 to 14.9]

4. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Flu A/CAL/7/09, Day 0 | 12
  Flu A/CAL/7/09, Day 21 | 48

5. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: as for outcome 4
Time Frame: At Days 0 and 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects for whom assay results for antibodies against A/California-like HA antigen for the blood sample taken 21 and 182 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Participants
  Flu A/CAL/7/09, Day 0 | 11
  Flu A/CAL/7/09, Day 182 | 40

6. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 Strain
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Titers
  Flu A/CAL/7/09, Day 0 | 6.6 [5.5 to 7.9]
  Flu A/CAL/7/09, Day 21 | 67.2 [46.1 to 98.0]

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 Strain
Description: as for outcome 6
Time Frame: At Days 0 and 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Titers
  Flu A/CAL/7/09, Day 0 | 6.5 [5.5 to 7.8]
  Flu A/CAL/7/09, Day 182 | 27.6 [19.2 to 39.8]

8. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: SCR was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Participants | 19

9. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Days 0 and 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Participants
  Flu A/CAL/7/09, Day 0 | 2
  Flu A/CAL/7/09, Day 182 | 21

10. Secondary Outcome: GMFR for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 3
Time Frame: At Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Fold change | 4.2 [3.0 to 6.0]

11. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:8 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/Netherlands/602/2009 (H1N1) (Flu A/Neth/602/09).
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects for whom assay results for antibodies against A/Netherlands-like HA antigen for the blood sample taken 21 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Flu A/Neth/602/09, Day 0 | 19
  Flu A/Neth/602/09, Day 21 | 41

12. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: as for outcome 11
Time Frame: At Days 0 and 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects for whom assay results for antibodies against A/Netherlands-like HA antigen for the blood sample taken 21 and 182 days after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Participants
  Flu A/Neth/602/09, Day 0 | 18
  Flu A/Neth/602/09, Day 182 | 41

13. Secondary Outcome: Titers for Neutralizing Antibodies Against Flu A/Netherlands/602/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:8. The flu strain assessed was Flu A/Netherlands/602/2009 (H1N1) (Flu A/Neth/602/09).
Time Frame: At Days 0 and 21
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Titers
  Flu A/Neth/602/09, Day 0 | 7.7 [5.8 to 10.1]
  Flu A/Neth/602/09, Day 21 | 29.3 [18.6 to 46.0]

14. Secondary Outcome: Titers for Neutralizing Antibodies Against Flu A/Netherlands/602/09 Strain of Influenza Disease
Description: as for outcome 13
Time Frame: At Days 0 and 182
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Titers
  Flu A/Neth/602/09, Day 0 | 7.5 [5.7 to 9.9]
  Flu A/Neth/602/09, Day 182 | 20.4 [14.4 to 28.7]

15. Secondary Outcome: Number of Subjects With Vaccine Response Rate (VRR) for Neutralizing Antibodies Against Flu A/Netherlands/602/09 Strain of Influenza Disease
Description: VRR for microneutralization titers was defined as the proportion of vaccinees with at least a 4-fold increase in post-vaccination reciprocal titer relative to Day 0. The flu strain assessed was Flu A/Netherlands/602/2009 (H1N1) (Flu A/Neth/602/09).
Time Frame: At Day 21
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 20

16. Secondary Outcome: Number of Subjects With VRR for Neutralizing Antibodies Against Flu A/Netherlands/602/2009 Strain of Influenza Disease
Description: as for outcome 15
Time Frame: At Day 182
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 49
Participants | 15

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Any Pain | 33
  Grade 3 Pain | 0
  Any Redness | 8
  Grade 3 Redness | 0
  Any Swelling | 5
  Grade 3 Swelling | 0

18. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Days
  Pain | 3.0 [2.0 to 4.0]
  Redness | 3.0 [1.5 to 6.0]
  Swelling | 2.0 [2.0 to 4.0]

19. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Headache, Joint pain at other location, Muscle aches, Shivering, Sweating and Fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0°C to ≤ 40.0°C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Any Fatigue | 10
  Grade 3 Fatigue | 1
  Related Fatigue | 9
  Any Headache | 7
  Grade 3 Headache | 1
  Related Headache | 7
  Any Joint pain | 1
  Grade 3 Joint pain | 0
  Related Joint pain | 1
  Any Muscle aches | 10
  Grade 3 Muscle aches | 0
  Related Muscle aches | 10
  Any Shivering | 2
  Grade 3 Shivering | 0
  Related Shivering | 2
  Any Sweating | 2
  Grade 3 Sweating | 0
  Related Sweating | 2
  Any Fever | 0
  Grade 3 Fever | 0
  Related Fever | 0

20. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Days
  Fatigue | 1.0 [1.0 to 3.0]
  Headache | 1.0 [1.0 to 3.0]
  Joint pain | 1.0 [1.0 to 1.0]
  Muscle aches | 3.0 [2.0 to 4.0]
  Sweating | 1.0 [1.0 to 1.0]
  Shivering | 1.0 [1.0 to 1.0]

21. Secondary Outcome: Number of Subjects With Medically Attended AEs (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 1

22. Secondary Outcome: Number of Subjects With MAEs
Description: as for outcome 21
Time Frame: During the 42-day (Days 0-41) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 7

23. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (from Day 0 up to Day 182)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 0

24. Secondary Outcome: Number of Subjects With Normal or Abnormal Hematological and Biochemical Levels
Description: Among hematological and biochemical parameters assessed were alanine aminotransferase (ALAT), albumin, alkaline phosphatase (AP), aspartate aminotransferase (ASAT), basophils, total bilirubin, bilirubin conjugated/direct, cholesterol, chloride, creatine, creatine kinase (CK), eosinophils, gamma-glutamyl transpeptidase (GGT), hematocrit, hemoglobin, potassium, lactate dyhydrogenase (LDH), lymphocytes, monocytes, sodium, neutrophils, platelets, protein, red blood cells, urate/uric acid, blood urea nitrogen (BUN) and white blood cells. Unknown = value unknown for the specified time point and laboratory parameter; Below = value below the laboratory reference range defined for the specified time point and laboratory parameter; Within = value within the laboratory reference range defined for the specified time point and laboratory parameter; Above = value above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Day 0 and Day 7
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  ALAT Unknown, Day 0 | 0
  ALAT Unknown, Day 7 | 0
  ALAT Below, Day 0 | 0
  ALAT Below, Day 7 | 0
  ALAT Within, Day 0 | 49
  ALAT Within, Day 7 | 50
  ALAT Above, Day 0 | 1
  ALAT Above, Day 7 | 0
  Albumin Unknown, Day 0 | 0
  Albumin Unknown, Day 7 | 0
  Albumin Below, Day 0 | 4
  Albumin Below, Day 7 | 6
  Albumin Within, Day 0 | 46
  Albumin Within, Day 7 | 44
  Albumin Above, Day 0 | 0
  Albumin Above, Day 7 | 0
  AP Unknown, Day 0 | 0
  AP Unknown, Day 7 | 0
  AP Below, Day 0 | 0
  AP Below, Day 7 | 0
  AP Within, Day 0 | 48
  AP Within, Day 7 | 48
  AP Above, Day 0 | 2
  AP Above, Day 7 | 2
  ASAT Unknown, Day 0 | 0
  ASAT Unknown, Day 7 | 0
  ASAT Below, Day 0 | 0
  ASAT Below, Day 7 | 0
  ASAT Within, Day 0 | 49
  ASAT Within, Day 7 | 50
  ASAT Above, Day 0 | 1
  ASAT Above, Day 7 | 0
  Basophils Unknown, Day 0 | 0
  Basophils Unknown, Day 7 | 0
  Basophils Below, Day 0 | 0
  Basophils Below, Day 7 | 0
  Basophils Within, Day 0 | 50
  Basophils Within, Day 7 | 49
  Basophils Above, Day 0 | 0
  Basophils Above, Day 7 | 1
  Total Bilirubin Unknown, Day 0 | 0
  Total Bilirubin Unknown, Day 7 | 0
  Total Bilirubin Below, Day 0 | 0
  Total Bilirubin Below, Day 7 | 0
  Total Bilirubin Within, Day 0 | 50
  Total Bilirubin Within, Day 7 | 50
  Total Bilirubin Above, Day 0 | 0
  Total Bilirubin Above, Day 7 | 0
  Bilirubin Conjugated/Direct Unknown, Day 0 | 0
  Bilirubin Conjugated/Direct Unknown, Day 7 | 0
  Bilirubin Conjugated/Direct Below, Day 0 | 0
  Bilirubin Conjugated/Direct Below, Day 7 | 0
  Bilirubin Conjugated/Direct Within, Day 0 | 50
  Bilirubin Conjugated/Direct Within, Day 7 | 50
  Bilirubin Conjugated/Direct Above, Day 0 | 0
  Bilirubin Conjugated/Direct Above, Day 7 | 0
  Cholesterol Unknown, Day 0 | 0
  Cholesterol Unknown, Day 7 | 0
  Cholesterol Below, Day 0 | 2
  Cholesterol Below, Day 7 | 2
  Cholesterol Within, Day 0 | 31
  Cholesterol Within, Day 7 | 36
  Cholesterol Above, Day 0 | 17
  Cholesterol Above, Day 7 | 12
  Chloride Unknown, Day 0 | 0
  Chloride Unknown, Day 7 | 0
  Chloride Below, Day 0 | 0
  Chloride Below, Day 7 | 0
  Chloride Within, Day 0 | 46
  Chloride Within, Day 7 | 44
  Chloride Above, Day 0 | 4
  Chloride Above, Day 7 | 6
  Creatine Unknown, Day 0 | 0
  Creatine Unknown, Day 7 | 0
  Creatine Below, Day 0 | 0
  Creatine Below, Day 7 | 1
  Creatine Within, Day 0 | 44
  Creatine Within, Day 7 | 43
  Creatine Above, Day 0 | 6
  Creatine Above, Day 7 | 6
  CK Unknown, Day 0 | 0
  CK Unknown, Day 7 | 0
  CK Below, Day 0 | 0
  CK Below, Day 7 | 1
  CK Within, Day 0 | 45
  CK Within, Day 7 | 43
  CK Above, Day 0 | 5
  CK Above, Day 7 | 6
  Eosinophils Unknown, Day 0 | 0
  Eosinophils Unknown, Day 7 | 0
  Eosinophils Below, Day 0 | 0
  Eosinophils Below, Day 7 | 0
  Eosinophils Within, Day 0 | 48
  Eosinophils Within, Day 7 | 48
  Eosinophils Above, Day 0 | 2
  Eosinophils Above, Day 7 | 2
  GGT Unknown, Day 0 | 0
  GGT Unknown, Day 7 | 0
  GGT Below, Day 0 | 0
  GGT Below, Day 7 | 0
  GGT Within, Day 0 | 41
  GGT Within, Day 7 | 41
  GGT Above, Day 0 | 9
  GGT Above, Day 7 | 9
  Hematocrit Unknown, Day 0 | 0
  Hematocrit Unknown, Day 7 | 0
  Hematocrit Below, Day 0 | 2
  Hematocrit Below, Day 7 | 3
  Hematocrit Within, Day 0 | 46
  Hematocrit Within, Day 7 | 47
  Hematocrit Above, Day 0 | 2
  Hematocrit Above, Day 7 | 0
  Hemoglobin Unknown, Day 0 | 0
  Hemoglobin Unknown, Day 7 | 0
  Hemoglobin Below, Day 0 | 7
  Hemoglobin Below, Day 7 | 8
  Hemoglobin Within, Day 0 | 43
  Hemoglobin Within, Day 7 | 42
  Hemoglobin Above, Day 0 | 0
  Hemoglobin Above, Day 7 | 0
  Potassium Unknown, Day 0 | 0
  Potassium Unknown, Day 7 | 0
  Potassium Below, Day 0 | 0
  Potassium Below, Day 7 | 1
  Potassium Within, Day 0 | 49
  Potassium Within, Day 7 | 48
  Potassium Above, Day 0 | 1
  Potassium Above, Day 7 | 1
  LDH Unknown, Day 0 | 0
  LDH Unknown, Day 7 | 0
  LDH Below, Day 0 | 0
  LDH Below, Day 7 | 1
  LDH Within, Day 0 | 50
  LDH Within, Day 7 | 49
  LDH Above, Day 0 | 0
  LDH Above, Day 7 | 0
  Lymphocytes Unknown, Day 0 | 0
  Lymphocytes Unknown, Day 7 | 0
  Lymphocytes Below, Day 0 | 1
  Lymphocytes Below, Day 7 | 0
  Lymphocytes Within, Day 0 | 49
  Lymphocytes Within, Day 7 | 50
  Lymphocytes Above, Day 0 | 0
  Lymphocytes Above, Day 7 | 0
  Monocytes Unknown, Day 0 | 0
  Monocytes Unknown, Day 7 | 0
  Monocytes Below, Day 0 | 0
  Monocytes Below, Day 7 | 0
  Monocytes Within, Day 0 | 47
  Monocytes Within, Day 7 | 47
  Monocytes Above, Day 0 | 3
  Monocytes Above, Day 7 | 3
  Sodium Unknown, Day 0 | 0
  Sodium Unknown, Day 7 | 0
  Sodium Below, Day 0 | 0
  Sodium Below, Day 7 | 0
  Sodium Within, Day 0 | 50
  Sodium Within, Day 7 | 50
  Sodium Above, Day 0 | 0
  Sodium Above, Day 7 | 0
  Neutrophils Unknown, Day 0 | 0
  Neutrophils Unknown, Day 7 | 0
  Neutrophils Below, Day 0 | 0
  Neutrophils Below, Day 7 | 1
  Neutrophils Within, Day 0 | 47
  Neutrophils Within, Day 7 | 49
  Neutrophils Above, Day 0 | 3
  Neutrophils Above, Day 7 | 0
  Platelets Unknown, Day 0 | 0
  Platelets Unknown, Day 7 | 1
  Platelets Below, Day 0 | 0
  Platelets Below, Day 7 | 1
  Platelets Within, Day 0 | 50
  Platelets Within, Day 7 | 48
  Platelets Above, Day 0 | 0
  Platelets Above, Day 7 | 0
  Protein Unknown, Day 0 | 0
  Protein Unknown, Day 7 | 0
  Protein Below, Day 0 | 2
  Protein Below, Day 7 | 3
  Protein Within, Day 0 | 45
  Protein Within, Day 7 | 46
  Protein Above, Day 0 | 3
  Protein Above, Day 7 | 1
  Red Blood Cells Unknown, Day 0 | 0
  Red Blood Cells Unknown, Day 7 | 0
  Red Blood Cells Below, Day 0 | 4
  Red Blood Cells Below, Day 7 | 4
  Red Blood Cells Within, Day 0 | 46
  Red Blood Cells Within, Day 7 | 46
  Red Blood Cells Above, Day 0 | 0
  Red Blood Cells Above, Day 7 | 0
  Urate/Uric acid Unknown, Day 0 | 0
  Urate/Uric acid Unknown, Day 7 | 0
  Urate/Uric acid Below, Day 0 | 1
  Urate/Uric acid Below, Day 7 | 1
  Urate/Uric acid Within, Day 0 | 45
  Urate/Uric acid Within, Day 7 | 45
  Urate/Uric acid Above, Day 0 | 4
  Urate/Uric acid Above, Day 7 | 4
  BUN Unknown, Day 0 | 0
  BUN Unknown, Day 7 | 0
  BUN Below, Day 0 | 0
  BUN Below, Day 7 | 0
  BUN Within, Day 0 | 44
  BUN Within, Day 7 | 44
  BUN Above, Day 0 | 6
  BUN Above, Day 7 | 6
  White Blood Cells Unknown, Day 0 | 0
  White Blood Cells Unknown, Day 7 | 0
  White Blood Cells Below, Day 0 | 2
  White Blood Cells Below, Day 7 | 2
  White Blood Cells Within, Day 0 | 46
  White Blood Cells Within, Day 7 | 48
  White Blood Cells Above, Day 0 | 2
  White Blood Cells Above, Day 7 | 0

25. Secondary Outcome: Number of Subjects With Abnormal Urine Sampling Parameters
Description: Among assessed urine sampling parameters were glucose, protein, red blood cells and urobilinogen.
Time Frame: At Day 0 and Day 7
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Glucose Negative, Day 0 | 49
  Glucose Positive, Day 0 | 1
  Glucose Negative, Day 7 | 45
  Glucose Positive, Day 7 | 5
  Protein Negative, Day 0 | 49
  Protein Positive, Day 0 | 1
  Protein Negative, Day 7 | 50
  Protein Positive, Day 7 | 0
  Red Blood Cells Negative, Day 0 | 45
  Red Blood Cells Positive, Day 0 | 5
  Red Blood Cells Negative, Day 7 | 43
  Red Blood Cells Positive, Day 7 | 7
  Urobilinogen Negative, Day 0 | 49
  Urobilinogen Positive, Day 0 | 1
  Urobilinogen Negative, Day 7 | 50
  Urobilinogen Positive, Day 7 | 0

26. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants
  Any AE(s) | 4
  Grade 3 AE(s) | 0
  Related AE(s) | 1

27. Secondary Outcome: Number of Subjects With Unsolicited AEs
Description: as for outcome 26
Time Frame: During the 42-day (Days 0-41) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Subjects
  Any AE(s) | 10
  Grade 3 AE(s) | 2
  Related AE(s) | 1

28. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 182)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix Group
Number analyzed (Participants) | 50
Participants | 4

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 42-day (Days 0-41) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 182).
Arm/Group | Arepanrix Group
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arepanrix Group (N=50)
Cataract (Eye disorders) | 1
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arepanrix Group (N=50)
Pain (General disorders) | 33
Redness (General disorders) | 8
Swelling (General disorders) | 5
Fatigue (General disorders) | 10
Headache (General disorders) | 7
Muscle aches (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.